CLINICAL TRIAL: NCT01903421
Title: Inhalational Anesthesia and Precipitation of Dementia: is There a Link? A Prospective, Multicenter, Randomized, Controlled Clinical Trial Comparing Two Different Anesthetic Techniques in Elderly Patients
Brief Title: Inhalational Anesthesia and Precipitation of Dementia: is There a Link?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-6122
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Elderly surgical patients; Alzheimer's disease; Dementia; Elderly; Surgery
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Fentanyl; Isoflurane; Sevoflurane; Hematologic Tests; Spinal Puncture; Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: The proposed study will be a prospective, multicenter, cluster randomization clinical trial comparing two different anesthetic techniques in elderly patients (> 65 years of age) undergoing urology/orthopedic/general surgery. The study will follow a cluster design; patients undergoing orthopedic or vascular surgery will have spinal anesthesia, where standard practice. Patients undergoing urology or general surgery will receive general anesthesia, also where it is standard practice. Patients with severe dementia will be excluded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia group (Active Comparator): Spinal anesthesia group will receive bupivacaine 10-15mg anesthesia according to the standard practice. Supplemental sedation with intravenous anesthetics (midazolam/propofol) will be optional.
  Interventions: Drug: Spinal anesthesia group: bupivacaine 10-15mg; Genetic: Blood test; Other: Lumbar spinal tap; Behavioral: Montreal Cognitive Assessment (MOCA) and MMSE
- General anesthesia group (Active Comparator): Induction of anesthesia will be achieved with propofol 1.5-2mg/kg and fentanyl 1-3g/kg. Anesthesia will be maintained with inhalational anesthesia (isoflurane or sevoflurane) at the discretion of anesthesiologist in charge of the case. A mixture of Air/O2 will be used to maintain adequate oxygenation. Nitrous oxide will not be used.
  Interventions: Drug: General anesthesia group: induction propofol 1.5-2mg/kg and fentanyl 1-3g/kg, maintained with isoflurane or sevoflurane; Genetic: Blood test; Other: Lumbar spinal tap; Behavioral: Montreal Cognitive Assessment (MOCA) and MMSE

INTERVENTIONS:
Drug: Spinal anesthesia group: bupivacaine 10-15mg
  Arms: Spinal anesthesia group
Drug: General anesthesia group: induction propofol 1.5-2mg/kg and fentanyl 1-3g/kg, maintained with isoflurane or sevoflurane
  Arms: General anesthesia group
Genetic: Blood test — DNA will be tested for the presence of ε4 allele of the apolipoprotein E gene
Other: Lumbar spinal tap — 1ml of cerebrospinal fluid (CSF) removed and stored for further analysis of amyloid tau protein after completion of the study
Behavioral: Montreal Cognitive Assessment (MOCA) and MMSE

SUMMARY:
Many elderly patients undergoing surgical procedures already have impaired cognitive (memory/concentration) status. Patients with pre-existing cognitive impairment, or dementia, may benefit from modified anesthesia techniques. It is estimated that one in eight people age 65 and older has Alzheimers disease. More so, nearly half of people that are 85 years or older have Alzheimers disease. Currently, both spinal (regional) and inhalational (general) anesthesia, are used in patients undergoing common urological, orthopedic, and general surgical procedures. Inhalational anesthesia has been associated with higher risk of memory impairment in experimental (animal) and human studies. However, currently, there are simply no large or good enough studies to be sure that inhalational anesthesia is responsible for causing dementia and Alzheimers disease.The proposed study investigates if elderly patients (65 years and older) undergoing spinal anesthesia (patient is awake or slightly sedated) are less likely to develop dementia and Alzheimers disease for up to 2 years after surgery, when compared to inhalational anesthesia (patient is kept asleep with gas anesthetic). The investigators will also test all patients for the presence of apolipoprotein (ApoE-Îμ4 type of gene that is present in 15-20% of patients), and beta-amyloid tau protein (present in cerebrospinal fluid) that are known risk factors for Alzheimers disease. The particular strength of this study is that it takes into account whether the frequency and/or severity of dementia and Alzheimers disease is different in patients with and without these markers. The investigators believe that this study will make a major contribution to better understanding of development of Alzheimers disease.

ELIGIBILITY:
Inclusion Criteria:

* >65 yrs of age
* Male or female
* Scheduled to undergo urologic procedures (e.g., transurethral resection of prostate, transurethral resection of bladder tumor), orthopedic (e.g., total knee replacement, total hip replacement) general (e.g., femoral hernia repair, lower abdominal surgery) or vascular surgery procedures (e.g. lower limb reperfusion amputations) and qualifies to be randomized to receive either local (spinal) or general anesthetic

Exclusion Criteria:

* Diagnosis of severe dementia
* Diagnosis of any other significant neurological disease such as Parkinson's, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain or spinal abnormalities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assessing the incidence of early dementia | Change from baseline, hospital discharge (3 day average), 3 months, 1 year, and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Djaiani, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (3):
- Canada (2):
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - William Osler Health Centre, Toronto, Ontario
- Pauls Stradins Clinical University Hospital, Riga, Latvia